CLINICAL TRIAL: NCT03384667
Title: Efficacy and Safety Evaluation of Maekmoondong-tang on Post-operative Cough in Patients With Lung Cancer -Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Maekmoondong-tang on Post-operative Cough in Patients With Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seong-Gyu Ko (Other)
Responsible Party: Sponsor-Investigator, Seong-Gyu Ko, Prof., Kyunghee University Medical Center
Organization: Kyunghee University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISEE_MMDT_2017
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Postoperative Cough; Lung Cancer
Keywords: Maekmoondong-tang; Mai-men-dong-tang; Bakumondo-to
MeSH Terms: conditions — Lung Neoplasms | interventions — maimendongtang

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMDT group (Experimental)
  Interventions: Drug: Maekmoondong-tang
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maekmoondong-tang — MMDT is a Herbal medicine consist of six herbs.
  Other Names: Maekgeuron Granules
  Arms: MMDT group
Drug: Placebo — The granules do not contain any active ingredients.
  Arms: Placebo group

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of Maekmoondong-tang on post-operative cough in patients with lung cancer. A randomized, double-blind, placebo-controlled trial will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years old.
* Patients undergone segmentectomy or lobectomy for lung cancer within 1 month
* Patients who do not or poorly respond to one week administration of common antitussive agents.
* Eastern Cooperative Oncology Group(ECOG) 0 to 2
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Patients undergoing adjuvant chemotherapy.
* Patients who have been diagnosed with acute respiratory disease within 1 month.
* Patients who have been diagnosed with bronchial asthma or bronchiectasis within 1 year
* Patients taking Angiotensin Converting Enzyme Inhibitor
* Patients with pseudoaldosteronism.
* Participants who have known prior hypersensitivity to any investigational product component
* Patient with acute or chronic infections requiring treatment (active HAV, HBV, HCV, HIV, TB)
* Pregnant or lactating females
* Women of childbearing potential
* Patient who do not agrees to use effective means of contraception and not to donate sperm during the trial and up to 1 month after final administration
* Patient who participated other clinical trials of medicine or medical devices within 1 month
* Individuals who are judged inappropriate for the study by investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Leicester Cough Questionnaire (LCQ) | Day 0 to Day 28
  Questionnaire used to measure quality of life in cough patients. The total score of LCQ is 3 to 21, and a higher score means a better quality of life.

SECONDARY OUTCOMES:
Cough VAS | Day 0 to Day 28
  Measure frequency and severity of cough by VAS
Yin deficiency scale | Day 0 to Day 28
  Questionnaire measures yin deficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea